CLINICAL TRIAL: NCT01858311
Title: Human Blood Outcomes Following Tocotrienol Supplementation - Nutrition Phase IIB NUTRITION PHASE IIB
Brief Title: Nutrition Blood Outcomes Following Tocotrienol N2B
Acronym: NIIB
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Collaborators: Malaysia Palm Oil Board (Other Government)
Responsible Party: Principal Investigator, Andrew Slivka, MD, Professor of Neurology, Ohio State University
Other Study IDs: 2012H0113
Record Dates: First submitted 2013-05-09; First posted 2013-05-21 (Estimated); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Stroke
Keywords: Stroke survivors; TIA survivors; Vitamin E; Carotech; Tocotrienol
MeSH Terms: conditions — Stroke | interventions — Tocotrienols

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood Draw
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Placebo vehicle: (2) placebo capsules following AM meal and (2) placebo capsules following PM meal.
  Interventions: Other: Placebo Vehicle
- Tocotrienol capsules (400 mg): (2) 100mg TCT capsules following AM meal and (2) 100mg TCT capsules following PM meal.
  Interventions: Dietary Supplement: Tocotrienol Capsules
- Tocotrienol Capsules (800 mg): (2) 200mg TCT capsules following AM meal and (2) 200mg TCT capsules following PM meal.
  Interventions: Dietary Supplement: Tocotrienol Capsules

INTERVENTIONS:
Dietary Supplement: Tocotrienol Capsules — Vitamin E TCT capsules- 400mg to 800mg per day (2 in the morning and 2 in the evening)
  Groups: Tocotrienol Capsules (800 mg); Tocotrienol capsules (400 mg)
Other: Placebo Vehicle — Placebo capsules per day (2 in the morning and 2 in the evening)
  Groups: Placebo vehicle

SUMMARY:
A natural form of vitamin E called tocotrienol (TCT) has blood thinning and cholesterol lowering properties, both of which may benefit stroke survivors. This study is being conducted to determine the blood thinning and cholesterol lowering properties of TCT in stroke or TIA (transient ischemic attack, which is also referred to as a "mini-stroke") survivors that are receiving the standard treatment for prevention of recurrent stroke.

Study Hypothesis: Oral TCT decreases the incidence of aspirin and clopidogrel nonresponders, increases the extent of inhibition of platelet aggregation, and decreases LDL without significant side effects in stroke patients.

DETAILED DESCRIPTION:
In this Phase IIB trial the goal is to determine the effects of orally supplemented TCT on platelet function and cholesterol as well as the safety in patients with TIA (transient ischemic attack) or stroke in addition to the standard treatment for stroke prevention. Recurrent cardiovascular events including stroke, TIA, heart attack, venous thrombosis, pulmonary embolism, systemic embolism will also be recorded. In patients with recurrent stroke, severity of the stroke and stroke size measured from MR (magnetic resonance) or CT (computed tomography) imaging will also be collected. We expect that TCT will inhibit blood clotting and lower cholesterol more than current standard treatment without significantly increasing bleeding risks or other side effects. Future work is planned in a larger TIA/stroke population to examine whether TCT adds to standard medical care in terms of decreasing incidence of stroke and improving outcomes following stroke.

ELIGIBILITY:
Inclusion Criteria:

* Patients with either atherothrombotic, cardioembolic, cryptogenic stroke or TIA (transient ischemic attack) for whom anticoagulation is not indicated
* Enrollment in trial must occur within 6 months of clinical presentation for first stroke or TIA event
* No history of long-term vitamin E supplement (defined as daily oral tocopherol or tocotrienol supplementation at least 6mos; within the past 5 years)
* No current vitamin E supplementation in multi-vitamin

Exclusion Criteria:

* Disabling stroke ( Modified Rankin Scale > 3)
* Prior intracranial hemorrhage (excluding traumatic)
* High risk of bleeding (recurrent gastrointestinal, genitourinary bleeding, active peptic ulcer disease)
* Anticipated requirement for long term use of anticoagulation
* Contraindications to antiplatelet agents (bleeding disorder, thrombocytopenia, prolonged INR)
* Irreversible medical condition likely to affect short-term survival or ability to participate in study such as cancer or other chronic disease with predicted survival of less than a year or severe psychiatric or neurologic disease that might complicate evaluation of study outcomes like dementia or schizophrenia
* Pregnancy or women of child bearing age who are not following an effective method of contraception
* Breast feeding
* Unable or unwilling to provide informed
* Unlikely to be compliant with therapy or unwilling to return for follow up frequent clinic visits
* Concurrent participation in another study with an investigational drug or devise
* Other likely specific cause of stroke such as dissection, infectious or noninfectious vasculitis, prothrombotic state

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Stroke survivors within 6 months of clinical presentation for ischemic stroke or TIA event
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2013-03; Primary Completion 2018-09 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
platelet aggregation activity | up to 1 year
  Platelet aggregation activity will be measured using standard clinical laboratory procedures

SECONDARY OUTCOMES:
Incidence of recurrent stroke | up to 1 year
  Incidence of recurrent stroke after previous diagnosed stroke or TIA.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - The Ohio State University, Columbus, Ohio
  - Mount Carmel Health System, Columbus, Ohio